CLINICAL TRIAL: NCT04539041
Title: A Randomized, Participant, Investigator and Sponsor Blinded, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Multiple Ascending Doses of Intrathecally Administered NIO752 in Participants With Progressive Supranuclear Palsy
Brief Title: Safety, Tolerability and Pharmacokinetics of Multiple Ascending Doses of NIO752 in Progressive Supranuclear Palsy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNIO752A02101
Record Dates: First submitted 2020-08-25; First posted 2020-09-04 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Progressive Supranuclear Palsy (PSP)
Keywords: progressive supranuclear palsy; PSP; antisense oligonucleotide; ASO; tau; NIO752; adult
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Pick Disease of the Brain | interventions — Oligonucleotides, Antisense

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort A NIO752 (Experimental): 4 injections of NIO752 at dose A
  Interventions: Drug: antisense oligonucleotide
- Cohort B NIO752 (Experimental): 4 injections of NIO752 at dose B
  Interventions: Drug: antisense oligonucleotide
- Placebo (Placebo Comparator): 4 injections of placebo
  Interventions: Drug: placebo
- Cohort C NIO752 (Experimental): 4 injections of NIO752 at dose C
  Interventions: Drug: antisense oligonucleotide
- Cohort D NIO752 (Experimental): 4 injections of NIO752 at dose D
  Interventions: Drug: antisense oligonucleotide
- Cohort E NIO752 (Experimental): 4 injections of NIO752 at dose E
  Interventions: Drug: antisense oligonucleotide

INTERVENTIONS:
Drug: antisense oligonucleotide — solution of antisense oligonucleotide injected intrathecally (spine tap) at multiple dose levels
  Other Names: NIO752
  Arms: Cohort A NIO752; Cohort B NIO752; Cohort C NIO752; Cohort D NIO752; Cohort E NIO752
Drug: placebo — placebo for each dose level
  Arms: Placebo

SUMMARY:
This is a phase 1, multi-center, double-blind, placebo-controlled, multiple dose escalation study with NIO752 in progressive supranuclear palsy (PSP) participants.

DETAILED DESCRIPTION:
This is a phase 1, multi-center, double-blind, placebo-controlled, multiple dose escalation study with NIO752 in progressive supranuclear palsy (PSP) participants.

Approximately 58 PSP participants in 5 cohorts will be randomized to receive NIO752 or placebo in a ratio of 3:1. Intrathecal (IT) injections will be given multiple times over 3 months and participants will remain in study for an additional 9-month follow-up period; or will be given multiple times over 9 months and participants will remain in study for an additional 3-month follow-up period.

Cohorts will be enrolled sequentially.

Safety assessments will include physical and neurological examinations, ECGs, vital signs, standard clinical laboratory evaluations (hematology, blood chemistry, and urinalysis), CSF laboratory test, adverse event, and serious adverse event monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Between 40 to 75 years old (inclusive)
3. Have PSP diagnosed for less than 5 years with a current classification of probable PSP Richardson syndrome, a progressive supranuclear palsy rating scale (PSPRS) score < 40 and MOCA score >17 at screening
4. Be able to ambulate independently or able to take at least 5 steps with minimal assistance
5. At least a 12-month history of postural instability or falls within 3 years from disease onset as per medical history
6. Vertical supranuclear gaze palsy, or reduced velocity of vertical saccade
7. Able and willing to meet all study requirements including:

   Have a study partner who is reliable, competent, and at least 18 years of age, and will be able to accompany the participant to study visits, be knowledgeable of the participant's ongoing condition during the study to provide study related information to study site when required both in person and via a phone Reside in a proximity to the study site to allow a timely unscheduled visit if necessary (ideally less than 2 hours) Able to undergo lumbar puncture (LP), CSF draws and blood draws
8. If the participant is receiving levodopa/carbidopa, levodopa/benserazide, a dopamine agonist, catechol-o-methyltransferase (COMT) inhibitor, rasagiline, CoQ10 or other Parkinson's medications, acetylcholinesterase inhibitors, antipsychotics, memantine, or other non-tau modifying Alzheimer's medication the dose must have been stable for at least 30 days prior to the screening visit and must remain stable for the duration of the study. No such medication can be initiated during the study.

Exclusion Criteria:

1. Live in a skilled nursing facility or dementia care facility
2. Evidence of motor neuron disease, or any other neurological disease that could explain symptoms
3. Clinically significant laboratory abnormality
4. Attempted suicide, suicidal ideation with a plan that required hospital admission within 12 months prior to Screening. In addition, patients deemed by the Investigator to be at significant risk of suicide, major depressive episode, psychosis, confusion state, or violent behavior should be excluded.
5. A clear and robust benefit from levodopa by history
6. Use of lithium, methylene blue or other putative disease modifying drugs for PSP within 30 days of screening
7. Any previous use of experimental therapy within 30 days or 5 half-lives prior to Day 1, whichever is greater
8. Any condition that increases risk of meningitis unless participant is receiving appropriate prophylactic treatment
9. History of post-lumbar-puncture headache of moderate or severe intensity and/or blood patch

11. Hospitalization for any major medical or surgical procedure involving general anesthesia within 12 weeks of Screening or planned during the study 12. Unable to undergo magnetic resonance imaging (MRI) due to for example claustrophobia, or presents absolute contraindications to MRI (e.g., metallic implants, metallic foreign bodies, pacemaker, defibrillator) 13. Patients with other significant brain MRI abnormalities by history or at screening.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Number of adverse events and serious adverse events | Baseline up to approximately one year (3-month treatment plus 9-month follow-up or 9-month treatment plus 3-month follow-up)
  Adverse events will be collected at clinical visits and other contacts. All abnormalities from safety assessments (physical exams and neurological exams and clinical safety labs) considered clinically significant will be recorded as adverse events
Change in severity scores for Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline up to approximately 1 year (3-month treatment plus 9-month follow-up or 9-month treatment plus 3-month follow-up)
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is a questionnaire that prospectively assesses Suicidal Ideation and Suicidal Behavior. The C-SSRS must be administered at visits. If, at any time after "screening and/or baseline" version, the score is "yes" on item 4 or item 5 of the Suicidal Ideation section of the C-SSRS or "yes" on any item of the Suicidal Behavior section, the participant must be referred to a mental health care professional for further assessment and/or treatment.
Levels of infection indicators in Cerebrospinal fluid (CSF) | Baseline up to approximately 1 year (3-month treatment plus 9-month follow-up or 9-month treatment plus 3-month follow-up)
  CSF safety labs measure levels of proteins, glucose, lactate and white blood cell counts with differential indicating infections.

SECONDARY OUTCOMES:
Concentrations of NIO752 in blood plasma | From the 1st dose administration (day 1), through study completion, where the longest duration would be approximately 1 year for those who receive 4 treatment doses
  concentrations of NIO752 in plasma
Concentrations of NIO752 in CSF | From the 1st dose administration (day 1), through study completion, where the longest duration would be approximately 1 year for those who receive 4 treatment doses
  concentrations of NIO752 in CSF
Cmax, Ctrough in blood plasma | From the 1st dose administration (day 1), through study completion, where the longest duration would be approximately 1 year for those who receive 4 treatment doses
  Maximum and trough level concentrations of NIO752 in plasma
Tmax in blood plasma | From the 1st dose administration (day 1), through study completion, where the longest duration would be approximately 1 year for those who receive 4 treatment doses
  Time of Cmax in plasma post first injection
AUClast in blood plasma | 0 to 24 hours after first injection
  Area under curve (AUC) from time zero to the last measurable concentration sampling time (tlast) (mass x time x volume-1)
AUCinf in blood plasma | 0 to 24 hours after first injection
  The AUC from time zero to infinity (mass x time x volume-1)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (3):
  - University of California San Diego, La Jolla, California
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Vanderbilt University Medical CenterX, Nashville, Tennessee
- Novartis Investigative Site, Montreal, Quebec, Canada
- Germany (6):
  - Novartis Investigative Site, Bonn, North Rhine-Westphalia
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
- Novartis Investigative Site, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to study results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18339
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2903